CLINICAL TRIAL: NCT05342844
Title: Comparison Between Two Different Doses of Dexmedetomidine as an Adjuvant to Bupivacaine in Ultrasound-guided Transversus Abdominis Plane Block for Postoperative Analgesia in Caesarean Delivery
Brief Title: Different Doses of Dexmedetomidine Added to Bupivacaine in Transversus Abdominis Plane Block in Caesarean Delivery
Acronym: TAP_dexmedet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, maha abou-zeid, Assistant Professor of Anesthesia and Surgical Intensive Care, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TAP-dexmedetomidine
Record Dates: First submitted 2022-04-11; First posted 2022-04-25 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: according to the computer-generated random number codes that will be placed in sealed envelopes, the patients will be randomly allocated into three groups; Group-Control, Group-Dexmedetomidine 0.5 and Group-Dexmedetomidine 1 according tho the local anesthetic injected in Ultrasound-guided bilateral Tranversus abdominis plane block
Who Masked: Participant, Investigator
Masking Description: The injectate used for TAPB will be prepared according to the group by an anesthesiologist who won't be involved in the data collection
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group-Control (No Intervention): After cession section, patients Will receive ultrasound (US)-guided bilateral transversus abdominis plane block with 10 mL bupivacaine 0.5% plus 10 mL normal saline 0.9% for each side
- Group-Dexmedetomidine 0.5 (Active Comparator): After cession section, patients Will receive ultrasound (US)-guided bilateral transversus abdominis plane block with 10 mL bupivacaine 0.5% plus 10 mL normal saline containing 0.5 mcg/kg dexmedetomidine for each side
  Interventions: Drug: Dexmedetomidine 0.5 mcg
- Group-Dexmedetomidine1 (Active Comparator): After cession section, patients Will receive ultrasound (US)-guided bilateral transversus abdominis plane block with 10 mL bupivacaine 0. 5% plus 10 mL normal saline containing 1 mcg/kg dexmedetomidine for each side
  Interventions: Drug: Dexmedetomidine 1 mcg

INTERVENTIONS:
Drug: Dexmedetomidine 0.5 mcg — 0.5 mcg/kg
  Arms: Group-Dexmedetomidine 0.5
Drug: Dexmedetomidine 1 mcg — 1 mcg/kg
  Arms: Group-Dexmedetomidine1

SUMMARY:
Cesarean birth is a common surgical procedure. After cesarean birth, postsurgical pain may delay recovery, interfere with maternal-newborn bonding, and reduce the breastfeeding if not adequately controlled. Postpartum analgesia has become a common concern.

Many adjuvant drugs used for peripheral nerve blocks as( N-methyl-d-aspartate (NMDA) receptor antagonists , Magnesium , Ephedrine , Dexamesathone , Fentanyl , Midazolam and Neostigmine) Dexmedetomidine is a potent and highly selective α2 adrenergic receptor agonist, exerts its sympatholytic effect by inhibiting the release of noradrenaline from central and peripheral sympathetic nerve endings. It is considered to be a useful agent with a wide safety margin, excellent sedative capacity and moderate analgesic properties

DETAILED DESCRIPTION:
This prospective double-blinded randomized controlled study will be done on parturients that are scheduled for elective cesarean delivery under spinal anesthesia to assess the efficacy of two different doses (0.5 mcg/kg and 1mcg/kg) of dexmedetomidine as an adjuvant to isobaric bupivacaine in TAPB compared to a control group on the postoperative analgesia in cesarean section under spinal anaesthesia

ELIGIBILITY:
Inclusion Criteria:

* Age from 19 to 40 years old
* American Society of Anesthesiologists (ASA) physical status II patients
* Singleton pregnancies with a gestational age of at least 37 weeks.
* Patients undergoing spinal anesthesia for cesarean delivery via a Pfannenstiel incision with exteriorization of the uterus.

Exclusion Criteria:

* Age < 19 or > 40 years.
* Height<150 cm, weight < 60 kg, body mass index (BMI) ≥40 kg/m2.
* Inability to comprehend or participate in the pain scoring system.
* Contraindications to spinal anesthesia (Coagulopathy, increased intracranial pressure, or local skin infection).
* Hypersensitivity to any drug used in the study.
* Any hypertensive disorders of pregnancy.
* Renal impairment or other contraindications to non-steroidal anti-infilamatory drugs (NSAIDS).
* Significant cardiovascular, renal or hepatic abnormalities.
* Patients with history of opioid intake, drug abusers or psychiatric patients

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — singleton pregnant women with a gestational age of at least 37 weeks
Enrollment: 81 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-14 (Actual)

PRIMARY OUTCOMES:
The time of the first postoperative analgesic requirement | during the first 24 postoperative hours

SECONDARY OUTCOMES:
Total amount of the postoperative analgesic drugs (ketolac, paracetamol and fentanyl) consumed in the | during the first 24 postoperative hours
  mg
The visual analog scale (VAS) scores during rest | during the first 24 postoperative hours
  11-point VAS (where 0 for no pain and 10 for the worst possible pain) at 0, 2, 4,6,12 and 24 hours postoperatively
The visual analog scale (VAS) scores during movement | during the first 24 postoperative hours
  11-point VAS (where 0 for no pain and 10 for the worst possible pain) at 0, 2, 4,6,12 and 24 hours postoperatively
Mean arterial blood pressure (MBP) | basal (preoperative), intraoperative each 10 minutes and postoperatively every hour during first 6 hours
  mmHg
heart rate (HR) | basal (preoperative), intraoperative each 10 minutes and postoperatively every hour during first 6 hours
  beat per minute
Patient satisfaction about the quality of postoperative analgesia | during the first 24 postoperative hours
  poor = 1, fair = 2, good = 3, excellent = 4
The side effects (nausea, vomiting, abdominal colic and lower limb weakness) | during the first 24 postoperative hours
  incidence
the time from intrathecal injection till regression of spinal anesthesia to L2 dermatome | during the first 24 postoperative hours
The level of sedation | during the first 24 postoperative hours
  using a 4-point scale (0 = awake and alert, 1 = minimally sedated, responds to speech, 2 = moderately sedated, arousable by tactile stimulation, and 3 = deeply sedated, arousable only by painful stimulation)

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University-Emergency hospital-ICU, Al Mansurah, Egypt